CLINICAL TRIAL: NCT05288777
Title: A Study of Adjuvant Chemoradiation and Biomarkers of Response in High-risk Breast Cancer
Brief Title: Adjuvant Chemoradiation and Biomarkers of Response in High-risk Breast Cancer
Acronym: Breast53
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Einsley-Marie Janowski, MD, Assistant Professor, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR210410
Record Dates: First submitted 2022-02-24; First posted 2022-03-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Radiation; Chemoradiation; Chemotherapy; Chemo; T-DM1; xeloda; capecitabine; Adjuvant; Combination treatment; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Capecitabine

STUDY DESIGN:
Intervention Model Description: Non-randomized assignment based on Her2/neu status and lymph node involvement
Who Masked: Outcomes Assessor
Masking Description: Participants, clinical research staff, and treating clinicians will be aware of arm assignment. The labels on research blood will not include the treatment arm on which the participant is assigned and this information will not be provided to lab investigators and staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Her2/neu positive and lymph node positive (Other): T-DM1/ trastuzumab emtansine infusion along with radiation to the breast or chest wall and lymph nodes
  Interventions: Drug: T-DM1; Radiation: External Beam Radiation Therapy 1
- Her2/neu positive and lymph node negative (Other): T-DM1/trastuzumab emtansine infusion along with radiation to the whole breast or chest wall
  Interventions: Drug: T-DM1; Radiation: External Beam Radiation Therapy 0
- Her2/neu negative and lymph node positive (Other): oral capecitabine twice per day along with radiation to the breast or chest wall and lymph nodes
  Interventions: Drug: Capecitabine; Radiation: External Beam Radiation Therapy 1
- Her2/neu negative and lymph node negative (Other): oral capecitabine twice per day along with radiation to the whole breast or chest wall
  Interventions: Drug: Capecitabine; Radiation: External Beam Radiation Therapy 0

INTERVENTIONS:
Drug: T-DM1 — Dosed at 3.6 mg/kg of body weight every 3 weeks for Her2/neu+ patients for a total duration of 14 cycles.
  Other Names: trastuzumab emtansine
  Arms: Her2/neu positive and lymph node negative; Her2/neu positive and lymph node positive
Drug: Capecitabine — Dosed at 825 mg/m2 +/- 150mg twice per day for a total duration of 6 months
  Other Names: xeloda
  Arms: Her2/neu negative and lymph node negative; Her2/neu negative and lymph node positive
Radiation: External Beam Radiation Therapy 0 — Dose of 40 Gy in 15 fractions to the whole breast or chest wall followed by consideration of a 10 Gy in 4 fraction boost to the lumpectomy cavity for a total duration of 15-19 days. Internal mammary nodal, dissected axilla coverage, and boost will be at the radiation oncologist's discretion.
  Other Names: EBRT
  Arms: Her2/neu negative and lymph node negative; Her2/neu positive and lymph node negative
Radiation: External Beam Radiation Therapy 1 — Dose of 40 Gy in 15 fractions to either the breast or chest wall along with comprehensive nodal radiation followed by consideration of a 10 Gy in 4 fraction boost for a total duration of 15-19 days. Internal mammary nodal, dissected axilla coverage, and boost will be at the radiation oncologist's discretion.
  Other Names: EBRT
  Arms: Her2/neu negative and lymph node positive; Her2/neu positive and lymph node positive

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of adjuvant chemoradiation therapy in high-risk breast cancer patients who had received neoadjuvant chemotherapy before their lumpectomy and/or mastectomy and were found to have residual disease. As well as examine the effects of this treatment combination on the immune system.

DETAILED DESCRIPTION:
Breast cancer is often treated with a combination of surgery, chemotherapy and radiation. In patients with advanced breast cancer, (neoadjuvant) chemotherapy is often given prior to surgical removal (lumpectomy and/or mastectomy). Neoadjuvant chemotherapy has been consistently shown to down-stage primary breast tumors and convert positive underarm lymph nodes to pathologically negative nodes. Residual disease discovered after receiving neoadjuvant chemotherapy indicates an increased risk for recurrence and poor overall survival. The combination of concurrent chemotherapy and radiation after surgery (adjuvant chemoradiation) may improve local and distant recurrence outcomes in high risk breast cancer patients. Chemoradiation is a standard treatment for many cancers and is universally associated with improvements in local recurrence, however, it has not historically been given as post-surgery breast cancer treatment.

The study will evaluate the safety, feasibility, and effectiveness of chemoradiation therapy in high-risk breast cancer patients. Radiation has been associated with various effects on immune cells. The study will also examine the effects of this combination on the immune cells.

Participants on this trial will be treated (per approved clinical guidelines) with capecitabine or Trastuzumab emtansine (T-DM1) depending on Her2 status while receiving radiation at the same time. Participants will have their blood drawn at various timepoints during treatment and follow up. Participants will also be asked to complete surveys asking about overall health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older
4. Diagnosis of stage I-IIIB breast cancer
5. Received neoadjuvant chemotherapy (minimum of 3 cycles) and surgical resection (lumpectomy and/or mastectomy)
6. Discovered to have residual disease at least ypT1aNx or ypTxN1mic at surgical resection
7. Candidate for adjuvant chemoradiation as part of standard clinical care
8. Planned initiation of radiation within 12 weeks of their final oncologic surgery
9. ECOG performance status ≤2
10. Adequate cardiac function, with LVEF greater or equal to 45% (only for patients who will receive TDM-1 therapy)
11. Adequate organ function per the following criteria within 21 days before the start of treatment. If a laboratory value required for study eligibility does not meet the below requirements, the value may be retested.

    * Absolute neutrophil count ≥1.5 k/uL
    * Platelets ≥100 k/uL
    * Hemoglobin ≥ 10 g/dL
    * Serum Creatinine ≤ 1.5 x ULN
    * Bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's disease, where bilirubin to 4x ULN is allowed).
    * AST and ALT ≤ 2.5 x ULN
    * Alkaline phosphatase ≤ 2.5 x ULN
12. For females and males of reproductive potential: agreement to use adequate contraception during study participation and for an additional 6 months after the end of chemoradiation administration or until advised by their medical oncologist
13. Agreement to adhere to Lifestyle Considerations throughout study duration
14. Subjects taking warfarin and plan to receive capecitabine will need their anticoagulant management assessed before starting treatment.

Exclusion Criteria:

1. Had a mastectomy with expander placement or immediate reconstructions
2. Diagnosed with systemic lupus
3. Diagnosed with scleroderma
4. Diagnosed with a genetic mutation associated with increased sensitivity to radiation (e.g. ataxia-telangectasias (AT)). AT heterozygotes without known radiation sensitivity may be included.
5. Acute bacterial or fungal infection requiring intravenous antibiotics at time of registration.
6. Pathologic evidence of metastatic disease, or strong clinical/radiological evidence of metastatic disease, at the investigator's judgment.
7. Pregnancy or lactation
8. Incarceration
9. Presence of cardiac pacemaker on side of the body that is being treated unless the pacemaker can be moved prior to treatment.
10. Anthracycline exposure exceeding a cumulative doxorubicin dose of 264 mg/m2 (240 mg/m2 plus a 10% threshold)
11. Known allergic reactions to components of capecitabine or T-DM1
12. Known DPD deficiency for patients prescribed capecitabine
13. Febrile illness within a week of starting treatment
14. Incomplete healing of chest wall or breast in the treatment field within 12 weeks from surgery.
15. Known HIV or active hepatitis.
16. Unwilling to discontinue endocrine therapy if currently taking endocrine therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Assess safety via toxicity grading | 1 year
  Assessment of toxicity frequency and severity using CTCAE v5.0 adverse event grading scale throughout chemoradiation treatment and follow up.
Assess feasibility via treatment delays and completion | 1 year
  Percent of participants completing adjuvant chemoradiation therapy and percent of participants requiring radiation or chemotherapy dose delays.

SECONDARY OUTCOMES:
Assess chronic cosmetic outcomes via LENT-SOMA scale | 1 year
  Assessment of chronic radiation-related cosmetic outcomes (e.g. dermatitis, telangiectasia, pigmentation, and radiation fibrosis) using "Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA)" scale throughout chemoradiation treatment and follow up. Each side effect is graded on a scale of 0 to 4, with higher scores meaning more severe outcome.
Assess acute cosmetic outcomes via RTOG/EORTC scale | 1 year
  Assessment of overall acute radiation related skin changes using the "Toxicity Criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC)" grading scale throughout chemoradiation treatment and follow up. Each side effect is graded on a scale of 0 to 4, with higher scores meaning more severe outcome.
Assess cosmetic outcomes via breast measurements | 1 year
  Measurement of breast tissue size by measuring tape/ruler.

OTHER OUTCOMES:
Estimate recurrence-free survival | 1 year
  Recurrence-free survival after 1 year of adjuvant chemoradiation therapy.
Describe the amount and type of immune cells via lab tests | 1 year
  Lab analysis (CBC w/ Differential and ELISA assays) of blood to characterize and count leukocyte populations (neutrophils, monocytes, lymphocytes) throughout adjuvant chemoradiation treatment and follow up.
Assess quality of life via RAND SF-36 patient survey | 1 year
  RAND SF-36 survey assesses feelings on overall health and activity level during follow up after adjuvant chemoradiation treatment.
Assess quality of life via FACT-B patient survey | 1 year
  Functional Assessment of Cancer Therapy- Breast (FACT-B) survey generally assess physical wellbeing, Social wellbeing, emotional wellbeing and functional well being during follow up after adjuvant chemoradiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Einsley Janowski, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No